CLINICAL TRIAL: NCT03068533
Title: The Use of 8% L-Arginine/Calcium Carbonate Containing Toothpaste in Comparison to Strontium Acetate Containing Toothpaste in Management of Hypersensitive Dentine in Chronic Periodontitis Patients : A Randomized-controlled Clinical Trial
Brief Title: 8% L-Arginine/Calcium Carbonate Toothpaste in Comparison to Strontium Acetate Toothpaste for Hypersensitive Dentin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdallah Hassan Mostafa, DR. Abdallah Hassan, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Abdallah Hassan
Record Dates: First submitted 2017-02-22; First posted 2017-03-03 (Actual); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Dentin Hypersensitivity
Keywords: DH, dentin hypersensitivity, chronic periodontitis
MeSH Terms: conditions — Dentin Sensitivity; Chronic Periodontitis | interventions — Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: similar empty tubes filled by the control and intervention toothpaste then sealed and given a number only.The patients,care provider,outcome assessor and investigator are blinded to the intervention and control toothpaste.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strontium acetate toothpaste (Active Comparator): All eligible patients will receive mechanical debridement in 1 or 2 sessions within 1 week before final evaluation.
  Interventions: Other: use of strontium acetate toothpaste
- Arginine/calcium carbonate toothpaste (Experimental): All eligible patients will receive mechanical debridement in 1 or 2 sessions within 1 week before final evaluation.
  Interventions: Other: 8% L-Arginine/calcium carbonate containing toothpaste

INTERVENTIONS:
Other: 8% L-Arginine/calcium carbonate containing toothpaste — use of 8% L-Arginine/calcium carbonate containing toothpaste to relieve hypersensitivity
  Arms: Arginine/calcium carbonate toothpaste
Other: use of strontium acetate toothpaste — use of strontium acetate toothpaste to relieve hypersensitivity
  Arms: Strontium acetate toothpaste

SUMMARY:
Dentinal hypersensitivity [DH] is a common condition in daily practice, especially in patients who have abrasion, attrition, gingival recession and erosion of teeth. It can affect individuals in the age range of 20-50 years.In a recent systematic review, it was reported that no gold standard treatment modality for dentin hypersensitivity has been established Thus there is a need to evaluate new formulations in different settings and in different populations and to compare those to commonly used agents seeking better results in pain relief for our patients. Studies showed that dentifrice formulations containing 8% arginine in combination with calcium carbonate and fluoride have the ability to plug dentinal tubules, by clumping of both arginine and calcium carbonate that bind with the negatively charged dentin . Aim of the study is to clinically evaluate toothpaste containing 8% arginine, calcium carbonate, and sodium mono-fluorophosphate, in comparison to toothpaste, containing 8% strontium acetate and NaF on the relief of DH in chronic periodontitis patients.

DETAILED DESCRIPTION:
1. Each eligible patient will be given a number.
2. All eligible patients will receive mechanical debridement in 1 or 2 sessions within 1 week before final evaluation.
3. The hypersensitive teeth will be isolated with cotton rolls, and stimuli will be applied to each tooth for final evaluation after scaling and debridement.
4. Air Sensitivity scale is used to assess sensitivity to air blast, while cold water test and tactile test will be held and assessed by Visual Analog Scale (VAS) , which score from 0 (no pain) to 10 (intense pain).
5. Patients will be handed a 30ml. white package written on it the previously assigned number to them and instructed to brush twice daily with the assigned toothpaste by a soft-bristled toothbrush for 8 weeks, with several returns to the clinic for re-evaluation and to take the refill of the assigned number of toothpaste.
6. Air blast sensitivity score and VAS will be evaluated again weekly and till the end of the evaluation period.

ELIGIBILITY:
Inclusion Criteria:

1. Slight to moderate chronic periodontitis patients diagnosed according to criteria of (Parameter on chronic periodontitis with slight to moderate loss of periodontal support.

   American Academy of Periodontology., 2000) as follows : Probing pocket depths up to 6mm Clinical attachment loss (CAL) up to 4mm Class I (incipient) furcation involvement Radiographic evidence of bone loss.
2. At least 2 teeth presenting hypersensitive areas on facial surfaces of teeth with score 2 or 3 on the air sensitivity scale (Pepelassi et al., 2015)
3. Provision of written informed consent

Exclusion Criteria:

1. Chipped teeth.
2. Defective restorations.
3. Deep dental caries or large restorations showing pulpal response.
4. Ongoing treatment with anti-inflammatory drugs.
5. Ongoing treatment for tooth hypersensitivity.
6. Pregnancy.
7. Uncontrolled metabolic diseases.
8. Psychiatric disorder.
9. Smoking

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-03-03 (Estimated); Study Completion 2018-04-01 (Estimated)

PRIMARY OUTCOMES:
change from baseline Pain (sensetivity) at 8 weeks | baseline and after 8 weeks
  This will be assessed using VAS that will be determined immediately before product use and then after 8 weeks of daily brushing with the test and control toothpastes following stimulus application using Visual Analog Scale (VAS)

SECONDARY OUTCOMES:
Probing pocket depth | baseline and after 8 weeks
  probing depth from gingival margin and till base of the pocket or sulcus in mm.
Gingival recession (GR) | baseline and after 8 weeks
  if present, distance between gingival margin to cemento-enamel junction in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Dr. Manal Hosni, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided